CLINICAL TRIAL: NCT01765881
Title: Comparison Between 25 µg Vaginal Misoprostol Versus Slow Release Pessary Prostaglandin-E2 (PGE2) : Could we Use Low Dose Vaginal Misoprostol as a First Line Treatment for Induction of Labor ?
Brief Title: Comparison Between 25 µg Vaginal Misoprostol vs Slow Release Pessary PGE2
Acronym: CYTOPRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1014301; 2011-000933-35 (EudraCT Number)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Delivery Uterine
Keywords: Induction of labor; cervical ripening; misoprostol,; prostaglandin; cost-effectiveness
MeSH Terms: interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Experimental): one 25 micrograms capsule all 4 hours by intravaginal route
  Interventions: Drug: Misoprostol
- Dinoprostone (Active Comparator): one unique intravaginal sustained released of 10 milligrams
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Drug: Misoprostol — administration of Misoprostol 25 micrograms capsule by intravaginal route every 4 hours, up to 4 capsules
  Other Names: CYTOTEC; 25 micrograms Misoprostol capsule by intravaginal route
  Arms: Misoprostol
Drug: Dinoprostone — administration of one sustained released pessary of 10 milligrams by intravaginal route
  Other Names: PROPESS; one intravaginal sustained released capsule of 10 milligrams
  Arms: Dinoprostone

SUMMARY:
For about 10% of pregnancies, it is necessary to induce delivery for medical reasons. Prostaglandins alone can be used to perform cervical ripening in cases of immature cervix. In France, dinoprostone is the own approved medication. It is in the form of gel or sustained release device whose effectiveness and side effects are comparable. The vaginal misoprostol has no marketing authorization in France, but is sometimes used. Some data in the scientific literature have showed that its use with low-dose (25 mcg) vaginally did not lead to more complications, was at least as effective and seems to be cost-effective compared with dinoprostone. Misoprostol with this dose and route of administration is now recommended by the American College of Obstetricians and Gynecologist (ACOG), Grade A (ACOG Practice Bulletin August 2009). This is not the case in France (French HAS 2008 Guidelines on induction of labor). According to HAS, the investigators still lack data on large samples to confirm the benefits of misoprostol 25 mcg vaginally, in terms of efficiency, rate of cesarean section, and lower cost compared to dinoprostone.

The primary objective is to demonstrate non-inferiority of vaginal misoprostol 25 mcg vs. dinoprostone in terms of cesarian section occurence with a non-inferiority margin of +5% difference.

DETAILED DESCRIPTION:
To show if the experimental treatment (25μg of intravaginal misoprostol) used for induction of labor in singleton women ≥ 36 weeks gestation with an unfavorable cervix is not clinically and statistically inferior than the reference treatment , ie intravaginal dinoprostone sustained release (10mg), in terms of cesarian sectionto compare the cost-effectiveness and to assess the differential tolerance of the two strategies.

Non-inferiority will be demonstrated if the upper limit of the 90%-bilateral confidence interval of the difference between cesarian section rates (misoprostol - dinosprostone) is below 5% in the intention-to-treat analysis and the per-protocol analysis.

If non-inferiority is demonstrated, as a secondary analysis, superiority of misosprostol will be tested.

Orther secondary objectives are to assess the cost-effectiveness, the tolerance, maternal satisfaction and other efficacy endpoints of the two strategies.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* Cephalic presentation
* Bishop ≤ 5
* ≤ 3 uterine contractions / 10 mn
* ≥ 36 weeks gestation
* Personally signed and dated informed consent document

Exclusion Criteria:

* History of cesarian-section
* uterine scar
* deceleration on Cardiotocogram (CTG)
* placenta praevia
* bleeding
* chorioamnionitis
* Fetal weight US ≥4500 g
* Contra-indication to vaginal delivery
* Hystory of myomectomy
* Herpes primoinfection or recurrence
* Allergy to prostaglandins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cesarean for all indications | Up to delivery
  Occurrence of cesarean section for all indications

SECONDARY OUTCOMES:
Cost-effectiveness of two strategies (direct medical cost differential efficiency strategies measured by the Cesarean rate | Up to discharge / end of study

OTHER OUTCOMES:
Adverse events | Up to discharge/end of study
  Summary description of all adverse events, related adverse events and serious adverse events by treatment using MedRA classification.
Other specific safety assessments | Up to discharge/end of study
  Maternal hyperstimulation syndromes with or without changes of foetal heart rate, uterine hypertonus, rate, rate of postpartum hemorrhage, degree III/IV perineal tears, uterine rupture, neonatal rate of pH <7.05 and/or BDbase deficit> 12mmol / L, rates Apgar score <7 at 5 minutes, transfer rate in neonatal intensive-care unit (NICU), neonatal seizures
Other efficacy assessments | Up to discharge/end of study
  Time from 1st treatment administration to delivery, ocytocine administration and dose, occurrence of instrumental delivery, occurrence of spontaneous delivery
Participant satisfaction assessment | Up to discharge/end of study
  Maternal satisfaction using visual analog scale and questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Vayssière, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - University Hospital Toulouse, Toulouse, France
  - Bicêtre Hospital, Le Kremlin-Bicêtre
  - Hospital Poissy, Poissy
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mounie M, Costa N, Gaudineau A, Molinier L, Vayssiere C, Derumeaux H. Cost-effectiveness analysis of vaginal misoprostol versus dinoprostone pessary: A non-inferiority large randomized controlled trial in France. Int J Gynaecol Obstet. 2022 Aug;158(2):390-397. doi: 10.1002/ijgo.13999. Epub 2021 Nov 19. PMID 34714938
- [Derived] Gaudineau A, Senat MV, Ehlinger V, Gallini A, Morin M, Olivier P, Roth E, Orusco E, Javoise S, Fort J, Lavergne C, Arnaud C, Rozenberg P, Vayssiere C; Groupe de Recherche en Obstetrique rt Gynecologie. Induction of labor at term with vaginal misoprostol or a prostaglandin E2 pessary: a noninferiority randomized controlled trial. Am J Obstet Gynecol. 2021 Nov;225(5):542.e1-542.e8. doi: 10.1016/j.ajog.2021.04.226. Epub 2021 Apr 19. PMID 33887241